CLINICAL TRIAL: NCT03368508
Title: Application of Photogrammetry for Manual Skills Training in Undergrad Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Technology (Other)
Responsible Party: Principal Investigator, Lo Chi Ngai, Principal Investigator, Singapore Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSS000001
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Healthy Individuals
Keywords: Simulation; Physiotherapy training; 360-degree video

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): the real-object rotatable 3D images were used in demonstrating these three techniques. The photogrammetry technique was used to produce the 3D images.
  Interventions: Behavioral: Simulating video
- Control group (Active Comparator): The control group received similar materials, but the only difference was that all the images were two-dimensional.
  Interventions: Behavioral: Conventional video

INTERVENTIONS:
Behavioral: Simulating video — A 360-degree simulating video showing physiotherapy assessment in lumbar area
  Arms: Experimental group
Behavioral: Conventional video — A conventional video showing physiotherapy assessment in lumbar area
  Arms: Control group

SUMMARY:
Education research shows that healthcare professional training can be made more efficient and effective with the integration of simulation technology. Despite the relevance of this technology in the training of medical students, evidence on its effectiveness in physiotherapy manual skills training is limited.

To compare the effectiveness of real-object three dimensional (3D) produced by Photogrammetry versus two dimensional (2D) images for the introduction of manual therapy skills to undergraduate physiotherapy students, with a blended learning activity.

DETAILED DESCRIPTION:
Using a randomised controlled trial design, first-year students enrolled in a 4-year bachelor with honours physiotherapy degree, participated in a 2-hour blended learning session. Three manual assessment techniques were presented - cervical compression, distraction and flexion-rotation tests. The techniques were demonstrated through two sets of learning materials with either real-object rotatable 3D images using Close-range Photogrammetry (experimental group) or traditional 2D computer images (control group). Students were examined after the training using an objective structured clinical evaluation (OSCE) procedure. The OSCE required the participants to demonstrate the three techniques learnt with the assessment criteria as therapist's position and skills, patient's position and overall management of the physical examination. The score of the standardized 9 item-practical performance test, with a maximum score of 54, was used as the primary outcome measure for analyses.

ELIGIBILITY:
Inclusion Criteria:

Physiotherapy students with no experience in spinal assessment

Exclusion Criteria:

People with unfavourable experience or responses to 360-degree video or VR/AR videos

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Structured objective clinical evaluation | Immediate
  Skills in assessment is assessed by a SOCE. The component evaluated skills in palpation, including: positioning of patient, direction of palpation contact, localization of specific structure, mobilization of segment during palpation, and precision of palpation.
  A nurmeric grading system (3 excellent, 0 incorrect) is used to assess each item.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Ngai Lo, Master, Principal Investigator — Singapore Institute of Technology
Locations (1):
- Singapore Institute of Technology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackstock FC, Jull GA. High-fidelity patient simulation in physiotherapy education. Aust J Physiother. 2007;53(1):3-5. doi: 10.1016/s0004-9514(07)70056-9. No abstract available. PMID 17326733
- [Background] Mori B, Carnahan H, Herold J. Use of Simulation Learning Experiences in Physical Therapy Entry-to-Practice Curricula: A Systematic Review. Physiother Can. 2015 Spring;67(2):194-202. doi: 10.3138/ptc.2014-40E. PMID 25931672
- [Background] Watson K, Wright A, Morris N, McMeeken J, Rivett D, Blackstock F, Jones A, Haines T, O'Connor V, Watson G, Peterson R, Jull G. Can simulation replace part of clinical time? Two parallel randomised controlled trials. Med Educ. 2012 Jul;46(7):657-67. doi: 10.1111/j.1365-2923.2012.04295.x. Epub 2012 May 30. PMID 22646319
- [Derived] Lo CN, Abdelkader T, Choi YM, Goff AJ, Suresh K, Carpio GAC, Soon B. Teaching Physiotherapy Students Physical Examination Skills by Using Photogrammetry: A Randomized Control Trial of 3- Versus 2-Dimensional Images. Simul Healthc. 2022 Feb 1;17(1):e98-e104. doi: 10.1097/SIH.0000000000000576. PMID 33867495